CLINICAL TRIAL: NCT03621488
Title: Randomized Controlled Study of the Efficacy of Behavioral Self-Activation Through Virtual Reality in the Treatment of Depression
Brief Title: Behavioral Self-activation and Virtual Reality in Depression
Acronym: DEPREVACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: C2care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL17_0215
Record Dates: First submitted 2018-07-25; First posted 2018-08-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Depression
Keywords: Behavioral Activation; Virtual reality; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of Behavioral Self-Activation with virtual reality (Experimental): 10 individual sessions of the Brief Behavioral Activation Treatment for Depression (BATD) program, lasting one hour, at the start of treatment, then half an hour thereafter, once a week
  + virtual reality activities of the session 4 to 9 lasting half an hour.
  Interventions: Other: Efficacy of Behavioral Self-Activation with virtual reality
- Efficacy of Behavioral Self-Activation without virtual reality (Sham Comparator): 10 individual sessions of the Brief Behavioral Activation Treatment for Depression (BATD) program, lasting one hour, at the start of treatment, then half an hour thereafter, once a week.
  Interventions: Other: Efficacy of Behavioral Self-Activation without virtual reality

INTERVENTIONS:
Other: Efficacy of Behavioral Self-Activation with virtual reality — Efficacy of Behavioral Self-Activation with virtual reality
  Arms: Efficacy of Behavioral Self-Activation with virtual reality
Other: Efficacy of Behavioral Self-Activation without virtual reality — Efficacy of Behavioral Self-Activation without virtual reality
  Arms: Efficacy of Behavioral Self-Activation without virtual reality

SUMMARY:
Depression is a major handicap in daily life and is often treated by behavioral activation (CA), including the Brief Behavioral Activation Treatment for Depression (BATD).The CA principle is to set up activities, in keeping with the values of the individual. Other tools associated with the CA deserve to be explored as virtual reality (VR), which offers scenarios and sensations similar to real life and a sense of life. in a safe and controlled environment, with the support of the therapist.The main objective is to compare the effectiveness of the program "BATD with RV" versus "BATD without RV" on the intensity of the depressive symptomatology and CA in everyday life.

Methodology: This is a randomized, blinded study. Inclusion criteria are: 18 to 70 years old; unipolar depression diagnosis; Showing a score of ≥ 17 on the BDI-II. 80 subjects will be recruited over 24 months and randomized into 2 groups: 1) intervention group program BATD in VR; 2) BATD program intervention group without RV, lasting 45 minutes.

Judgment Criteria: The effectiveness of the intervention will be evaluated by the BDI-II scale and the Behavioral Activation for Depression Scale (BADS).

Outcomes: A new management of depression (AC with RV) to improve the quality of life of the patient; proof of its effectiveness; a generalization of this care; and recognition of its effectiveness in the scientific community.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 70,
2. Having a diagnosis of unipolar depressive disorder characterized (diagnostic criteria of depression of DSM-V),
3. Primary depression and not secondary to another disorder (eg social phobia, OCD, severe personality disorder, ASD, TCA, ect.)
4. Showing a score greater than or equal to 17 points on the IDB-II,
5. Followed by a psychiatrist from the University Hospital of Montpellier or a liberal,
6. Can read, understand and speak French,
7. To be affiliated or beneficiary of a social security scheme.
8. Collection of informed consent.

Exclusion Criteria:

(1) History of head trauma or recent central neurological conditions only (2) Current treatment by seismotherapy or rTMS or CBT. (3) Exclusion from all substance-related disorders except tobacco-related disorder (DSM-V)

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Evolution of depression | 0 and 6 months
  Beck Depression Inventory version II (BDI-II; depression) ; decrease BDI-II score between 0 and 6 months.

SECONDARY OUTCOMES:
Evolution of depressive symptoms | 0, 3 and 6 months
  Inventory of Depressive Symptomatology by the clinician (IDS-C) ; decrease IDS-C score between 0 and 3 months ; and between 0 and 6 months.
Evolution of depression | 0 and 3 months
  Beck Depression Inventory version II (BDI-II; depression) ; decrease BDI-II score between 0 and 3 months.
Life quality | 3 and 6 months
  The Short Form (36) Health Survey (SF36) ; increase quality of life in the end of the treatment and three months later.
Physical fatigue | 3 and 6 months
  Multidimensional Fatigue Inventory (physical fatigue); Reduce the level of physical fatigue, in the end of the treatment and three months later.
Number of activities | 3 and 6 months
  Number of spontaneous activities performed during the week. Increase the number of activites in daily life in the end of the treatment and three months later.
Hopelessness | 3 and 6 months
  Beck Hopelessness scale (feelings about the future, loss of motivation, and expectations); increase hope, in the end of the treatment and three months later.
Therapeutic alliance | 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 weeks; 13 and 6 months
  Attendance at sessions and visits during all the study.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine CAPDEVIELLE, MD, PhD, Study Director — University Hospitals of Montpellier, France
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No